CLINICAL TRIAL: NCT05870358
Title: Melatonin Supports Non Surgical Periodontal Treatment in Patients With Type 2 Diabetes and Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yağmur Saraç Gül (Other)
Responsible Party: Sponsor-Investigator, Yağmur Saraç Gül, One of the principal investigator, Recep Tayyip Erdogan University
Organization: Recep Tayyip Erdogan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RecepTayyipErdoganU.2
Record Dates: First submitted 2023-03-25; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Periodontitis; Melatonin; Matrix Metalloproteinases
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fmSRP (No Intervention): 27 patients with diabetic periodontitis underwent full mouth scaling and root planning (fmSRP) alone
- fmSRP-mel (Active Comparator): 28 patients with diabetic periodontitis were administered systemic melatonin tablets (6 mg daily, for 30 days) immediately after fmSRP.
  Interventions: Drug: Melatonin 3 MG

INTERVENTIONS:
Drug: Melatonin 3 MG — In this clinical trial, all patients that have both diabetes mellitus and periodontitis were performed full mouth scaling and root planning in order to start their periodontal treatments. Different from the control group, in fmSRP-mel group's patients systemic melatonin tablets (6 mg daily, for 30 days) were given immediately after the fmSRP procedure in order to support the scaling and root planning.
  Other Names: Melatonina 3mg
  Arms: fmSRP-mel

SUMMARY:
Background and aim: Hyperinflammatory host response associated with diabetes mellitus significantly provokes periodontal tissue destruction. In this context, supporting the standard treatment of periodontitis in diabetics with host modulation agents is a current field of study.

This clinical study aims to investigate the clinical efficacy of melatonin supplementation in non-surgical periodontal treatment in patients with Type 2 DM and periodontitis and its biological basis (clinical effectiveness) based on some basic markers.

Material and method: In this randomized controlled and double-blind study, 27 of 55 patients with diabetic periodontitis underwent full mouth scaling and root planning (fmSRP) alone and 28 of them were administered melatonin (6 mg daily, for 30 days) in addition to fmSRP. The possible therapeutic contribution of melatonin was evaluated clinically and biochemically [gingival crevicular fluid (GCF) RANKL, OPG and MMP-8 and serum IL-1β levels] at 3 and 6 months.

DETAILED DESCRIPTION:
Ethical Approval This double-blind and randomized controlled clinical study was carried out on 55 patients with Type 2 DM and periodontitis who applied to the Periodontology Clinic of the Faculty of Dentistry of Recep Tayyip Erdoğan University between 2021/February and 2022/January and met the study criteria. Ethical approval was given by the Clinical Research Ethics Committee of the Faculty of Medicine of the same university within the framework of the Declaration of Helsinki (2008) (2022/03). The possible risks and benefits of the treatment to be applied to the participants were mentioned and their verbal and written consents were obtained.

Working Groups According to the WHO, in individuals in the young age category, "stage 3/4 periodontitis" was determined according to the current periodontal disease and condition classification as the diagnostic criterion for periodontitis. Accordingly, probing pocket depth (PPD) should be at least 6mm and bone loss should be at least 3mm. Our diagnostic criteria for Type 2 DM was fasting plasma glucose (FPG) level greater than 126 mg/dl and glycosylated hemoglobin level (HbA1c) greater than 6.5%. Those who smoke, use antibiotics, anti-inflammatory and antioxidant drugs in the last 6 months, work night shifts, are in pregnancy and lactation, have cancer and autoimmune diseases, have kidney disease, have received any periodontal treatment in the last 6 months obese patients were also excluded from the study. In Europe, obesity is defined as a body-mass index (BMI) of more than 30 kg/m2 and a waist circumference of more than 88 cm in women and 102 cm in men.

Treatment Protocol According to the above criteria, patients included in the study were randomly divided into control (fmSRP) and treatment [fmSRP-melatonin (fmSRP-mel)] groups by a computer program by an independent researcher (HA). The investigator (YSG), who provided the sample and conducted the clinical procedures, was blind to the study groups. fmSRP is the approach of completing supragingival and subgingival debridement procedures within 24 hours with periodontal curettes, scalers and ultrasonic instruments. Additional melatonin administration was made in the form of tablets containing 6mg of melatonin daily for 30 days from the day following the SRP. Patients were instructed to take the tablets just before bedtime. No additional application was made in the control group. Within the scope of the non-surgical periodontal treatment program, all patients were trained on brushing teeth with the modified bass technique and the use of appropriate interface cleaning tools. These trainings were repeated in the maintenance sessions. Participants were also instructed not to use any mouthwash.

Sample Collection and Clinical Periodontal Measurements Clinical periodontal measurements with gingival crevicular fluid(GCF) and serum samples were performed at baseline (T0) and at 3th (T1) and 6th months (T2) following fmSRP. In all three periods, sampling was done one day before clinical periodontal measurements.

GCF samples were taken from the interproximal regions of the two teeth with the most radiographic bone loss in each of the four quadrants in the morning. Initially, proper isolation was achieved by means of cotton rolls. The area was slightly dried for 10 seconds. Sterile paper strips (Periopaper, Proflow, Inc., Amityviile, NY) were advanced until minimal resistance was felt in the sulcus. Waited 30 seconds. Paper strips contaminated with blood or saliva were not included. The GCF volume in each paper strip was measured using the periotron device (Periotron 8010 Harco Electronics, Winnipeg, Canada) by electrical compedance method and recorded as µl. Immediately afterwards, 8 paper strips obtained from each patient were transferred to an eppendorf tube containing 250 µl of phosphate buffer solution. It was stored in a -80°C freezer (Thermo Fisher Scientific, Waltham, MA, USA) until the day of biochemical analysis.

Immediately following the GCF samples, 16 cc venous blood samples were taken from the left arm antecubital fossa region of the patients. After the blood was centrifuged at 3000 rpm at 2-8oC for 15 minutes, serum samples were obtained (Elektro-mag, Istanbul, Turkey). The samples were taken into Eppendorf tubes and kept in a -80°C freezer (Thermo Fisher Scientific, Waltham, MA, USA) until the day of analysis.

Plaque index (PI), gingival index (GI), bleeding on probing (BOP), PPD and clinical attachment level (CAL) measurements were performed for clinical periodontal status assessments. PPD was measured as the distance between the deepest point of the sulcus and the gingival margin, and CAL as the distance between the deepest point of the sulcus and the enamel-cementum junction. Scoring for each tooth was made from 6 different regions for PPD and CAL, and from 4 different regions for other indices. Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) was used for measurements.

Biochemical Analysis Eppendorf tubes, which were removed from the freezer 24 hours before the experiment, were allowed to thaw gradually, first at -20oC and then at +4oC. The samples and reagents were brought to room temperature (18-25oC) just before the analysis. RANKL (Catalog no: E-EL-H5813), OPG (Catalog no: E-EL-H1341) and MMP-8 (Catalog no: E-EL-H1450) analyzes in GCF samples, IL-1ß (Catalog no: E- EL-H0149) analyzes were performed on serum samples using the enzyme-linked immunosorbent assay (ELISA) method and according to the instructions of the kit manufacturer (Elabscience, Houston, Texas, USA). Results were calculated as ng/ml (MMP-8) and pg/ml (IL-1β, RANKL and OPG).

Statistical Analysis Windows 17.0 for SPSS program was used for statistical analysis. (SPSS Inc., Chicago, USA) The conformity of the data to the normal distribution was evaluated with the Shapiro Wilk test. The Mann Whitney U test was used for intergroup comparisons, and the Friedman, Wilxocon tests and Bonferroni correction were used for the analysis of time-dependent within-group changes. Chi-square test was applied for comparison between groups in terms of genders. A p<0.05 level was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* According to the WHO, in individuals in the young age category (18-65 years)
* Periodontitis diagnosed patients, "stage 3/4 periodontitis" was determined according to the current periodontal disease and condition classification as the diagnostic criterion for periodontitis
* Diabetic patients, our diagnostic criteria for Type 2 DM was fasting plasma glucose level greater than 126 mg/dl and glycosylated hemoglobin level (HbA1c) greater than 6.5%.

Exclusion Criteria:

* Smoke, use antibiotics, anti-inflammatory and antioxidant drugs in the last 6 months
* Work night shifts
* Pregnancy and lactation
* Cancer and autoimmune diseases
* Kidney disease
* Periodontal treatment in the last 6 months
* Obese patients (In Europe, obesity is defined as a body-mass index of more than 30 kg/m2 and a waist circumference of more than 88 cm in women and 102 cm in men)

Ages: 31 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Clinical Findings: Plaque index score(PI) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  According to the tooth Plaque index, each tooth surface was divided into 4 separate regions and the plaque intensity for each region is scored as:
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
  Finally, scores are collected and calculate the arithmetic mean for the mouth score.
Clinical Findings: Gingival index score (GI) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  The criteria are entirely confined to qualitative changes in the gingival soft tissue.Periodontal probe was used and gently inserted the sulcus. Each tooth surface was divided into 4 separate regions and the gingival bleeding activity for each region is scored as:
  0 = Normal gingiva
  1. = Mild inflammation -slight change in color, slight oedema. No bleeding on probing
  2. = Moderate inflammation-redness, oedema and glazing. Bleeding on probing
  3. =Severe inflammation -marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
  Finally, scores are collected and calculate the arithmetic mean for the mouth score.
Clinical Findings: Bleeding on probing(BOP) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  Each tooth surface was divided into 4 separate regions and gently probed by using periodontal probe.There is a bleeding as a positive score, and there is no bleeding as a negative score. The BOP is considered positive if bleeding occurred between 30 seconds after probing. Whole the probed area and positive score area ratio were calculated and BOP(%)score was found.
Clinical Findings:Probing pocket depth (PPD) | Change from baseline(T0) to 3rd month (T1) and 6th month (T2)
  Probing pocket depth (PPD) measured with a periodontal probe on 6 different points around each tooth. PPD is known as distance between gingival margin and the base of the pocket/sulcus. By using periodontal probe(Williams periodontal probe) 6 different points are measured. Each scores of surfaces are collected and averaged for the mouth score for PPD.
Clinical Findings: Clinical Attachment Level (CAL) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  By using periodontal probe(Williams periodontal probe) 6 different points are measured.CAL, distance from the bottom of the pocket to the cemento-enamel junction of tooth. If there is gingival recession, recession depth is also added the CAL. By using periodontal probe(Williams periodontal probe) 6 different points are measured. Each scores of surfaces are collected and averaged for the mouth score for CAL.
Biochemical Findings: RANKL (pg/ml) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  RANKL (pg/ml) were measured samples from gingival crevicular fluid by using commercial ELİSA kits according to the instructions of the kit manufacturer
Biochemical Findings: OPG (pg/ml) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  OPG (pg/ml) were measured samples from gingival crevicular fluid by using commercial ELİSA kits according to the instructions of the kit manufacturer
Biochemical Findings: MMP-8(ng/ml) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  MMP-8(ng/ml) were measured samples from gingival crevicular fluid by using commercial ELİSA kits according to the instructions of the kit manufacturer
Biochemical Findings: IL-beta(pg/ml) | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  IL-beta(pg/ml) were measured samples from serum by using commercial ELİSA kits according to the instructions of the kit manufacturer
Biochemical Findings: RANKL/OPG | Change from baseline(T0) to 3rd month(T1) and 6th month(T2)
  RANKL/OPG, numeric ratio that can be indicated as only numeric value(no need some kind of units)

CONTACTS AND LOCATIONS:
Locations (1):
- Yagmur Sarac Gul, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No